CLINICAL TRIAL: NCT05427630
Title: Inhaled Cannabis Versus Placebo for the Acute Treatment of Migraine: a Pilot, Randomized, Double-blind, Placebo-controlled, Crossover, Dose-ranging Trial
Brief Title: Dose-Ranging Trial of Inhaled Cannabis for Acute Migraine Treatment
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate funding
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Nathaniel Schuster, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 802999
Record Dates: First submitted 2022-06-17; First posted 2022-06-22 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Migraine; Cannabis; THC
Keywords: Migraine; Cannabis; THC
MeSH Terms: conditions — Migraine Disorders; Marijuana Abuse | interventions — Dronabinol; nabiximols; THC 5; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled, Dose-ranging Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each participant will have an identification number and randomization of drug sequence allocation will be performed a priori using a random number generator by the study pharmacist. The 4 treatments will be identically encapsulated by the study pharmacist. The study pharmacist will place the capsules in identical sealed plastic bags labeled "Migraine 1" through "Migraine 4."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- THC ~2.5% (Experimental): Inhalation of cannabis flower containing THC ~2.5%
  Interventions: Drug: THC ~2.5%
- THC ~5% (Experimental): Inhalation of cannabis flower containing THC ~5%
  Interventions: Drug: THC ~5%
- THC ~10% (Experimental): Inhalation of cannabis flower containing THC ~10%
  Interventions: Drug: THC ~10%
- Sham Cannabis (Sham Comparator): Inhalation of cannabis flower from which the THC and CBD have been extracted
  Interventions: Drug: Sham Cannabis

INTERVENTIONS:
Drug: THC ~2.5% — Cannabis flower containing THC ~2.5%
  Other Names: THC; delta 9-tetrahydrocannabinol; marijuana
  Arms: THC ~2.5%
Drug: THC ~5% — Cannabis flower containing THC ~5%
  Other Names: THC; delta 9-tetrahydrocannabinol; marijuana
  Arms: THC ~5%
Drug: THC ~10% — Cannabis flower containing THC ~5%
  Other Names: THC; delta 9-tetrahydrocannabinol; marijuana
  Arms: THC ~10%
Drug: Sham Cannabis — Cannabis flower from which the THC and CBD have been extracted
  Other Names: Placebo; Sham
  Arms: Sham Cannabis

SUMMARY:
This pilot crossover study will evaluate 3 different potencies of inhaled cannabis (2.5%, 5%, and 10%) and inhaled placebo cannabis for the acute treatment of migraine.

DETAILED DESCRIPTION:
In this double-blind, randomized, crossover trial, subjects will treat 4 separate migraine attacks with 4 different treatments. Inhaled cannabis will be administered using a portable system. Subjects will self-administer inhaled cannabis as early as possible in the course of a migraine, taking 4 puffs of 1) THC 2.5%, 2) THC 5%, 3) THC 10%, or 4) placebo. Patients will treat each of the 4 distinct migraine attacks with a different cannabis sample. Outcomes measured will include pain freedom, most bothersome symptom (MBS), and pain relief as well as presence or absence of photophobia, phonophobia, and nausea at 15 minutes, 30 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 24 hours, and 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 and ≤ 65
* Able to communicate in English
* Migraine, with or without aura, in its episodic or chronic manifestations, as per the International Headache Society (IHS) classification International Classification of Headache Disorders (ICHD-3) criteria (section 1.1, 1.2, 1.3).(48)
* Ability to provide informed consent and complete website questionnaires in English
* Agrees not to use cannabis outside of the study during participation in the study
* Agrees not to use opioids or barbiturates during participation in the study
* Agrees not to drive a motor vehicle within 4.5 hours following last use of inhaled cannabis during participation in the study

Exclusion Criteria:

* Positive urine drug test for THC, barbiturates, opioids, oxycodone, or methadone prior to enrollment
* Pregnancy
* Breastfeeding
* Prisoner
* Known cognitive impairment
* Institutionalized
* Current moderate-severe or severe depression
* Current or past history of bipolar depression, schizophrenia, or psychosis
* Current or past history of cannabis, alcohol, opioid, or amphetamine abuse or other substance use disorder at the discretion of the research team
* Active pulmonary disease, class IV heart failure, cirrhosis, or other severe medical illnesses at the discretion of the research team.
* Allergy to cannabis

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Headache Pain Freedom at 2 Hour Post-Treatment | 2 Hours Post-Treatment
  Dichotomous outcome of pain freedom defined as reduction from moderate/severe pain to no pain

SECONDARY OUTCOMES:
Most Bothersome Symptom (MBS) Freedom at 2 Hours Post-Treatment | 2 Hours Post-Treatment
  Dichotomous outcome of resolution of most bothersome symptom (of photophobia, phonophobia, or nausea) selected at the beginning of the migraine prior to cannabis administration
Headache Pain Relief at 2 Hours Post-Treatment | 2 Hours Post-Treatment
  Dichotomous outcome of pain reduction defined as reduction from moderate/severe pain to mild/no pain

OTHER OUTCOMES:
Headache pain freedom | 15 minutes, 30 minutes, 1 hour, 1.5 hours, 4 hours, 24 hours, 48 hours
  Dichotomous outcome of reduction from moderate/severe to no pain
Most bothersome symptom (MBS) | 15 minutes, 30 minutes, 1 hour, 1.5 hours, 4 hours, 24 hours, 48 hours
  Dichotomous outcome of resolution of MBS (of photophobia, phonophobia, or nausea) selected at the beginning of the migraine prior to cannabis administration
Headache pain relief | 15 minutes, 30 minutes, 1 hour, 1.5 hours, 4 hours, 24 hours, 48 hours
  Dichotomous outcome of reduction from moderate/severe to mild/no pain
Freedom from photophobia | 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 24 hours, 48 hours
  Dichotomous outcome of resolution of photophobia
Freedom from phonophobia | 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 24 hours, 48 hours
  Dichotomous outcome of resolution of phonophobia
Freedom from nausea | 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 24 hours, 48 hours
  Dichotomous outcome of resolution of nausea
Freedom from vomiting | At any time over 48 hours
  Dichotomous outcome of whether patient vomited during this migraine attack
Use of rescue medication | At any time over 48 hours
  Dichotomous outcome of use of rescue medication
Sustained pain freedom | 24 hours and 48 hours
  Dichotomous outcome of absence of headache pain at 2 hours after dose, with no use of rescue medication and no recurrence of headache pain
Sustained most bothersome symptom freedom (MBS) | 24 hours and 48 hours
  Dichotomous outcome of absence of MBS at 2 hours after dose, with no use of rescue medication and no recurrence of MBS

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel M Schuster, MD, Principal Investigator — Center for Pain Medicine, UC San Diego
Locations (1):
- Center for Pain Medicine, UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared in a manner TBD based on funding availability and journal requirements
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 1 year and ending 5 years after article publication
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be sent to nmschuster@health.ucsd.edu